CLINICAL TRIAL: NCT03968146
Title: Ultrasound Guided Erector Spinae Plane Block in Scoliotic Adolescents Undergoing Posterior Spine Instrumentation . A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block in Scoliotic Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, maged gamal, anethesia demonstrator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-15-2019
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence; Erector Spinae Plane Block
MeSH Terms: conditions — Scoliosis | interventions — Fentanyl; Neoadjuvant Therapy; Maintenance; Morphine; Meperidine; Ketorolac; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): patients will receive Erector Spinae plane block in addition to intravenous fentanyl
  Interventions: Procedure: Erector Spinae Plane Block; Drug: Fentanyl; Drug: rescue Morphine; Drug: pethidine; Drug: Ketorolac; Drug: Acetaminophen
- Group C (Other): Control group will receive only intravenous fentanyl.
  Interventions: Drug: Fentanyl; Drug: additional Fentanyl; Drug: Morphine; Drug: rescue Morphine; Drug: pethidine; Drug: Ketorolac; Drug: Acetaminophen

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The linear multi-frequency 6-13 megahertz transducer will be used. In the prone position,under aseptic conditions, the probe will be placed in a longitudinal position 2-3 cm lateral to the vertebral column. The transverse processes of the vertebrae at (mid) level of surgery, the Erector Spinae muscle and the psoas muscle are identified. A 22 gauge echogenic needle will be inserted in an in plane technique in a cephalad to caudad direction until bone contact with the top of the transverse process is reached. After slight retraction of the needle, A test dose of 5% dextrose in water can expand the fascial plane and confirm needle-tip location prior to injection of local anaesthetic. Then, 0.5 ml/kg of bupivacaine 0.25% with 0.1 mg/kg dexamethasone and adrenaline 1 : 200000 will be injected between erector spinea muscle and transverse process, taking in consideration not exceeding the toxic dose of bupivacaine; 4 mg/kg . the same procedure will be repeated on the contralateral side.
  Arms: Group E
Drug: Fentanyl — patients will receive an induction dose at 1 mcg/kg. If the analgesia was inadequate in the form of increase in heart rate and or arterial blood pressure by more than 20% of baseline values during surgery, this warrants the administration of intravenous fentanyl (0.5µg/kg).
  Other Names: fentanyl for induction and maintenance
Drug: additional Fentanyl — patients will receive another dose of fentanyl 1 µg/kg 1 minute before start of skin incision.
  Arms: Group C
Drug: Morphine — After end of surgery and emergence from anesthesia, patients will receive continuous intravenous morphine with 0.03 mg/kg/hr.
  Other Names: morphine infusion
  Arms: Group C
Drug: rescue Morphine — Morphine IV will be given as rescue analgesia (20 µg/kg) in all study groups if VAS pain score more than 3. The total maximum hourly morphine is 0.75 mg/kg/hr.
Drug: pethidine — After reaching maximum hourly morphine and the patient is still in pain, pethidine will be used as a rescue at 0.5 mg/kg.
Drug: Ketorolac — patients will receive IV ketorolac from the postoperative second day 15 mg q 6 hours, not to exceed 5 days.
Drug: Acetaminophen — patients will receive postoperative IV acetaminophen IV 10 mg/ kg q 6 hours

SUMMARY:
For scoliotic surgeries, Erector Spinae Plane Block (ESPB) can add to the multimodal approach for perioperative pain management with decreasing the opioids requirement, improving recovery and decreasing ICU stay.

DETAILED DESCRIPTION:
All patients will be assessed clinically and investigated for Pulmonary function test and Echocardiography. Laboratory work needed will be: Complete blood count (CBC); prothrombin time and concentration (PT& PC); partial thromboplastin time (PTT); bleeding time (BT); clotting time (CT) and liver function tests.

an online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into the two study groups. Random allocation numbers will be concealed in opaque closed envelops.participants and those assessing/analyzing the outcome(s) will be blind to group assignment.

Eutectic Mixture of Local Anesthetics (EMLA) cream will be applied to the site of venous puncture. After insertion of venous access, all children will receive midazolam at a dose of 0.1 mg/Kg. Intraoperative monitoring will include continuous electrocardiogram (ECG), pulse oximetry, invasive arterial blood pressure, end-tidal carbon dioxide (CO2), inhaled gas analyzer and temperature monitoring.

General anesthesia will be induced in both groups (Erector Spinae group and control group) using propofol 2.5 mg/kg over 20-30 seconds, atracurium 0.5 mg/kg to facilitate endotracheal intubation and fentanyl 1 µg/kg. Anesthesia will be maintained using isoflurane (1 MAC) and atracurium infused as 0.5 mg/kg/hr. All patients will receive IV ranitidine 2 mg/kg, ondansetron 0.1 mg/kg, cefotaxime 50 mg/kg and acetaminophen 15 mg/kg. An arterial catheter and a urinary catheter will be placed. Then patients will be turned to the prone position.

In group E: will receive Erector Spinae Plane Block (ESPB) In group C: control group will receive another dose of fentanyl 1 µg/kg 1 minute before start of skin incision. After end of surgery and emergence from anesthesia, patients will receive continuous intravenous morphine with 0.03 mg/kg/hr.

In both groups, if the analgesia obtained from both methods of ESBP or IV fentanyl was inadequate in the form of increase in heart rate and or arterial blood pressure by more than 20% of baseline values during surgery, this warrants the administration of intravenous fentanyl (0.5µg/kg). Total blood loss, duration of surgery, number of vertebral levels fixed, total fentanyl consumed will be recorded. After completion of surgical procedure and emergence from anesthesia the patient will be referred to post-anaesthesia care unit (PACU). Quality of analgesia will be assessed immediately postoperative and then at 4, 8, 12, 16, and 24 hours postoperatively in the Intensive Care Unit (ICU) by using VAS pain score. All patients will receive postoperative IV acetaminophen IV 10 mg/ kg q 6 hours, ketorolac from second day 15 mg q 6 hours, not to exceed 5 days. Patients will also receive ranitidine 2 mg/kg q 12 hours. Vital signs and urinary output will be monitored. Morphine IV will be given as rescue analgesia (20 µg/kg) in all study groups if visual analogue scale (VAS) pain score more than 3. The total maximum hourly morphine is 0.75 mg/kg/hr. After reaching maximum hourly morphine and the patient is still in pain, pethidine will be used as a rescue at 0.5 mg/kg. Morphine will be stopped if maximum hourly dose is reached or the patient becomes sedated (Ramsay score >2), has a ventilatory rate of <12 bpm, or an oxygen saturation of <95%, or has a serious adverse event (allergy, hypotension, severe vomiting).

Patients will be continuously monitored in the PACU and ICU. Naloxone and full resuscitation equipment are available. Time of first need for morphine and total 24 hr morphine consumption will be recorded. Complications e.g nausea, vomiting, pruritis or respiratory depression will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesia classification (ASA) I-II
* Patients undergoing dorsal spine instrumentation for scoliosis.

Exclusion Criteria:

* Refusal of block.
* Bleeding tendency with prothrombin concentration PC less than 75 % or platelet count less than 150,000/µL.
* Skin lesion, wounds or infection at the puncture site.
* Known allergy to local anaesthetic drugs.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | the first 24 hours post-operative period.
  Total postoperative rescue morphine consumption in mg/kg for each group in the first 24 hours post-operative period.

SECONDARY OUTCOMES:
Total fentanyl consumption | intraoperative period
  Total intraoperative fentanyl consumption in mcg/kg for each group.
Visual Analogue Scale | the first 24 hours post-operative period.
  the visual analogue scale (VAS) is for Pain assessment It is a * total 10 cm * linear scale for pain it ranges from minimum ( 0 for no pain at all ) to maximum ( 10 for the worst pain imaginable ) higher number values indicate worst outcome. For example, as the patient mark the scale nearer to maximum, this indicate more severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided